CLINICAL TRIAL: NCT01138618
Title: Hematological Clozapine Monitoring With a Point-of-care Device (CHEMPAQ)
Acronym: CHEMPAQ
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aalborg Psychiatric Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1.5 - 01 MARCH2010
Record Dates: First submitted 2010-05-21; First posted 2010-06-07 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2011-11

CONDITIONS: Schizophrenia
Keywords: Clozapine; hematological monitoring; CHEMPAQ; Granulocytes; WBC
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CHEMPAQ-venous-CHEMPAQ-venous: The two arms only differ in order of kind of blood samples.
  Interventions: Device: Venous blod sample; Device: CHEMPAQ
- Venous-CHEMPAQ-Venous-CHEMPAQ: The two arms only differ in order of kind of blood samples.
  Interventions: Device: Venous blod sample; Device: CHEMPAQ

INTERVENTIONS:
Device: Venous blod sample — Regular venous blood sample withdrawn from the laboratory
Device: CHEMPAQ — Capillary blood sample analyzed by CHEMPAQ

SUMMARY:
Clozapine remain the drug of choice for treatment resistant schizophrenia and up to 60% of patients not responding to other antipsychotics will respond to clozapine. However, the use of clozapine is restricted due to the risk of agranulocytosis and consequently the need for mandatory hematological monitoring. CHEMPAQ XBC is a point-of-care device that can be used in patients home and analyze WBC and granulocytes by a single capillary blood drop. This study aims to investigate whether this new procedure increases the acceptability of clozapine

ELIGIBILITY:
Inclusion Criteria:

* Treated with clozapine
* Compliant with blood monitoring
* Willing to give informed consent

Exclusion Criteria:

* Prior case of agranulocytosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with clozapine
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Pain sensation | Monthly for four months
  Pain sensation was measured using a visual analog scale (VAS)

SECONDARY OUTCOMES:
The benefits of CHEMPAQ | Monthly for four months
  Caregivers and patients were asked about the benefits of using CHEMPAQ for hematological clozapine monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Jimmi Nielsen, MD, Principal Investigator — Aalborg Psychiatric Hospital, Aarhus University Hospital
Locations (6):
- Denmark (6):
  - Psychiatric Center Roskilde, Greve, Greve
  - Aalborg Psychiatric Hospital, Aalborg
  - Psychiatric Center Aarhus, Aarhus
  - Psychiatric Center Copenhagen, Copenhagen
  - Psychiatric Centre Esbjerg, Esbjerg
  - Psychiatric Center Odense, Odense

REFERENCES:
- [Background] Kane J, Honigfeld G, Singer J, Meltzer H. Clozapine for the treatment-resistant schizophrenic. A double-blind comparison with chlorpromazine. Arch Gen Psychiatry. 1988 Sep;45(9):789-96. doi: 10.1001/archpsyc.1988.01800330013001. PMID 3046553